CLINICAL TRIAL: NCT03745196
Title: A Double-blind, Placebo-controlled Study to Assess the Effects of Inhaled PC945 in the Treatment of Culture-positive Aspergillus or Candida Fungal Bronchitis in Subjects With Moderate to Severe Asthma or Other Chronic Respiratory Diseases.
Brief Title: The Effect of PC945 on Aspergillus or Candida Lung Infections in Patients With Asthma or Chronic Respiratory Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is being terminated early as a result of the coronavirus (COVID-19) outbreak.
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC_ASP_004; 2018-000244-26 (EudraCT Number)
Record Dates: First submitted 2018-10-24; First posted 2018-11-19 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Asthma; Respiratory Candidiasis; Respiratory Aspergillosis; COPD; Bronchiectasis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC945 (Experimental): PC945 5mg once-daily, nebulized
  Interventions: Drug: PC945
- Placebo (Placebo Comparator): Placebo, nebulized
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PC945 — Study drug under investigation
  Arms: PC945
Drug: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
This study tests the effects of an experimental drug PC945 in people with asthma or other chronic respiratory diseases whose lungs are infected by Aspergillus fungi and Candida yeasts.

PC945 may be useful in treating patients infected with Aspergillus as, unlike the usual treatments, it is inhaled into the lung and has been designed to stay there and treat the infection. Participants will continue to receive their usual treatment for their chronic respiratory disease. Half of the participants will receive PC945 and half will receive a placebo. The amount of fungus and yeast in the patients' phlegm will be measured over the course of the study. The study will take place at multiple sites in UK and will include approximately 46 participants. The maximum study duration will be about 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be male or female, aged 18 years (inclusive) or older (at the time of consent).
2. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose and requirements of the study and is willing to participate.
3. Subject's diagnosis of moderate to severe asthma (GINA Step 3 or 4) made by a respiratory physician and treated with an inhaled steroid or other chronic respiratory disease.

   1. For subjects with asthma, the diagnosis of asthma must be supported either by:

      * i. Historical evidence of:

        * 1. Increased airway hyper-responsiveness (methacholine PC20 <8 mg/ml).
        * or
        * 2. Airflow obstruction (FEV1/FVC ratio of less than 70%) and short-term variations in FEV1 (>12%).
      * or
      * ii. Bronchodilator reversibility ≥12% or ≥200 mL improvement in FEV1 post bronchodilator after administration of a short-acting beta agonist at screening.

      OR
   2. Subjects with other chronic respiratory disease (such as COPD or bronchiectasis) susceptible to fungal bronchitis.
4. Subject must have a positive sputum fungal culture with one or more colonies of A. fumigatus complex / A. niger complex or 200 or more colonies of yeast measured using a modified standard approach on one occasion obtained within the 28-day screening period.
5. Subject must be able to produce a spontaneous sputum sample.

Exclusion Criteria:

1. Subjects who have received more than 2 weeks of intravenous (IV), oral or inhaled antifungal therapy within 6 months prior to Visit 3 or any antifungal therapy (IV, oral or inhaled) within 2 months of Visit 3.
2. Subjects taking medication that could significantly increase the risks of AEs with triazoles.
3. Subjects who are receiving antiretroviral protease inhibitors.
4. Clinical or laboratory evidence of bacterial bronchitis at the point of screening.
5. Subjects who have used an experimental medical device or received an experimental drug within 3 months or within a period less than five times the experimental drug's half-life, whichever is longer, before the first dose of the study drug is scheduled.
6. Clinically significant screening abnormalities (including, but not limited to, vital signs, ECG, laboratory tests, physical examination and spirometry) that, in the Investigator's opinion, exclude the subject from participation in the study.
7. Positive test at screening for hepatitis B virus infection, or antibodies to hepatitis C virus.
8. If female, the subject is pregnant (e.g. has a positive serum β human chorionic gonadotropin at screening or a positive urinary pregnancy test pre-dose on Day 1), lactating or breast feeding.
9. Subject is an employee or a first-degree relative of anyone employed by Pulmocide, a participating clinical trial site, or any contract research organisation involved in the study.
10. Any other reason that the Investigator considers makes the subject unsuitable to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of Aspergillus fumigatus (A. fumigatus) complex / Aspergillus niger (A. niger) complex colonies on sputum culture | Baseline to Day 32-35
  This is a binary endpoint
Reduction in the numbed of colonies of Candida species (spp) on sputum culture | Baseline to Day 32-35
  Substantial reduction in colony forming unit (CFU) count by at least 50%

SECONDARY OUTCOMES:
Predicted post bronchodilator forced expiratory volume in 1 second (FEV1) values | Baseline to Day 84
Forced vital capacity (FVC) values | Baseline to Day 84
The number of sputum A. fumigatus complex / A. niger complex CFUs in fungal culture | Baseline to Day 84
Sputum A. fumigatus measured by quantitative polymerase chain reaction (qPCR) | Baseline to Day 84
Spontaneous sputum weight (24-hour collection) | Baseline to Day 84
The number of sputum Candida spp. CFUs in fungal culture | Baseline to Day 84
C. albicans measured by qPCR in sputum | Baseline to Day 84
The concentration of A. fumigatus-specific immunoglobulin G (IgG) as measured in serum | Baseline to Day 84
Serum Total immunoglobulin E (IgE) levels | Baseline to Day 84
A. fumigatus-specific IgE levels | Baseline to Day 84
Change in Asthma control questionnaire - 6 item [ACQ6] (Total score) in asthma patients only | Baseline to Day 84
Change in Asthma Quality of Life Questionnaire - Juniper [AQLQ-J] (Total score) in asthma patients only | Baseline to Day 84
Change in St George's Respiratory Questionnaire [SGRQ] (Total score) | Baseline to Day 84
Change in Leicester Cough Questionnaire (Total score) | Baseline to Day 84
Breathlessness visual analogue scale rating, change over time | Baseline to Day 84
  Symptom severity rated from "Best ever" to "Worst possible"
Correlation between A. fumigatus measured by qPCR and clinical response | Baseline to Day 84
Correlation between Candida albicans measured by qPCR and clinical response | Baseline to Day 84
Area undertake curve from time 0 to 2h post dose (AUC(0-2)) | Baseline to Day 84
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
Last quantifiable plasma concentration (Ct) | Baseline to Day 84
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
maximum observed concentration (Cmax) | Baseline to Day 84
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
concentration at the end of the dosage interval (Ctrough) | Baseline to Day 84
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
Adverse events (AEs) incidence (safety and tolerability) | Baseline to Day 84
Twelve-lead electrocardiogram (ECG) (Safety parameter) | Baseline to Day 84
  including QT interval corrected for Bazetts formula, QT interval, QRS Interval, PR Interval and ventricular rate).
Proportion of participants who meet the markedly abnormal criteria for vital signs assessment at lease once post dose | Baseline to Day 84
Proportion of participants who meet the markedly abnormal criteria for safety laboratory assessment at lease once post dose | Baseline to Day 84
Change in peak expiratory flow rate [PEFR] | Baseline to Day 84
Antibiotic use | Baseline to Day 84
Sputum characteristics - consistency and presence of blood (fresh morning sputum samples) | Baseline to Day 84
Sputum colour (fresh morning sputum samples) | Baseline to Day 84

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Glenfield Hospital, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Royal Brompton Hospital, London
  - Northwest Lung Research Centre, Manchester